CLINICAL TRIAL: NCT02488993
Title: PROSPER: Prospective Real World Outcomes Study of Hepatic Encephalopathy Patients' Experience on Rifaximin-α (TARGAXAN®/XIFAXAN®) 550 mg
Brief Title: Real World Outcomes Study of Hepatic Encephalopathy Patients' Experience on Rifaximin (PROSPER)
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Other Study IDs: ZZ2014GL03
Record Dates: First submitted 2015-06-15; First posted 2015-07-02 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prospective Phase Rifaximin-α 550mg: Prospective data collection of patients treated with Rifaximin-α 550mg from point of study entry.
  Interventions: Other: Prospective Phase Rifaximin-α 550mg
- Prospective Phase No Rifaximin-α 550mg: Prospective data collection of patients NOT treated with Rifaximin-α 550mg from point of study entry.
  Interventions: Other: Prospective Phase No Rifaximin-α 550mg
- Retrospective Phase: Review of medical records and electronic hospital admissions data for patients with HE who have not received Rifaximin-α 550mg within the previous 12 months.
  Interventions: Other: Retrospective Phase

INTERVENTIONS:
Other: Prospective Phase Rifaximin-α 550mg — Prospective data collection of all patients receiving rifaximin-α 550 mg from the point of study entry.
  Other Names: TARGAXAN; XIFAXAN
  Groups: Prospective Phase Rifaximin-α 550mg
Other: Prospective Phase No Rifaximin-α 550mg — Prospective data collection of all patients not receiving rifaximin-α 550 mg from the point of study entry.
  Groups: Prospective Phase No Rifaximin-α 550mg
Other: Retrospective Phase — Review of medical records and electronic hospital admissions data for patients with HE who have not received rifaximin-α 550 mg during the previous 12 months.
  Groups: Retrospective Phase

SUMMARY:
This study evaluates hepatic encephalopathy (HE) and liver-related hospitalization rates and duration of stay in patients with HE treated with rifaximin-α 550mg compared to patients receiving other therapies.

This registry study aims to comprehensively and rigorously characterize the impact of rifaximin-α 550 mg on hospitalization, clinical safety and effectiveness outcomes, and quality of life in patients with HE in Europe and Australasia.

DETAILED DESCRIPTION:
Whilst clinical trial data and a few small observational studies have demonstrated the potential of rifaximin-α 550 mg to reduce overt HE episodes and hospitalizations, there is a need by physicians, commissioners and other healthcare professionals caring for patients with HE to understand the impact of management with rifaximin-α 550 mg on healthcare resource use in real world clinical practice. Currently available data are from evaluations undertaken in single UK centres. In addition, the overall burden of HE has not been well characterized, including the impact on patient quality of life, or impaired productivity incurred by patients' caregivers. This multinational, multicentre disease registry study aims to comprehensively and rigorously characterize the impact of rifaximin-α 550 mg on hospitalization, clinical safety and effectiveness outcomes, and quality of life in patients with HE in Europe and Australasia. The study will expand upon previous work in the following ways:

* Provide characterization of the burden of HE and the impact of rifaximin-α 550 mg in a real world setting, to complement RCT evidence;
* Allow for more rigorous characterization of the impact of rifaximin-α 550 mg on patient outcomes for individuals with HE over time. This will be achieved by prospectively enrolling patients not taking rifaximin-α 550 mg to characterize outcomes over time in the absence of treatment, and by assessing the quality of life and workplace productivity implications of HE.

There will be no change to the management of patients for the purposes of this study beyond normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis;
* Patient is ≥18 years of age;
* Patient is enrolled within 12 weeks of resolution of an episode of overt HE associated with a hospital visit;
* Patient is able to provide informed consent to participate in the study (individually or via caregiver);
* Patient meets clinical eligibility to receive rifaximin-α 550 mg in the opinion of the participating physician, regardless of HE treatment actually received.

Exclusion Criteria:

* West Haven Conn score of ≥2 at time of study entry (i.e. at provision of informed consent);
* Mental health disorder such as dementia or psychosis which makes diagnoses of HE questionable;
* Prior treatment with rifaximin in the 12 months before qualifying episode of overt HE associated with a hospital visit;
* Contraindications to the use of rifaximin-α as per local summary of product characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis aged 18 years or over who are enrolled within 12 weeks of resolution of an episode of overt HE associated with a hospital visit, who are eligible for treatment with rifaximin-α 550 mg.
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2015-06; Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
HE and liver related hospitalization rate in patients receiving rifaximin- α 550mg compared to other therapies | 12 months

SECONDARY OUTCOMES:
All-cause hospitalization rate in patients with HE receiving rifaximin-α 550 mg compared to those receiving other therapies | 12 months
Global Evaluation of Treatment Effectiveness of rifaximin-α 550 mg compared to other therapies | 12 months
Chronic Liver Disease Questionnaire (CLDQ) to evaluate effectiveness of rifaximin-α 550 mg compared to other therapies | 12 months
Number of sublects with adverse events after rifaximin-α 550 mg compared with other therapies | 12 months
Work productivity and Activity Impairment Questionnaire to evaluate quality of life in patients with HE | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ng, Study Director — Norgine
Locations (1):
- Queen Elizabeth Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Krag A, Schuchmann M, Sodatonou H, Pilot J, Whitehouse J, Strasser SI, Hudson M. Design of the Prospective Real-world Outcomes Study of hepatic encephalopathy Patients' Experience on Rifaximin-alpha (PROSPER): an observational study among 550 patients. Hepatol Med Policy. 2018 Jan 8;3:4. doi: 10.1186/s41124-017-0029-9. eCollection 2018. PMID 30288327